CLINICAL TRIAL: NCT02864992
Title: A Phase II Single-arm Trial to Investigate Tepotinib in Advanced (Locally Advanced or Metastatic) Non-small Cell Lung Cancer With METex14 Skipping Alterations or MET Amplification (VISION)
Brief Title: Tepotinib Phase II in NSCLC Harboring MET Alterations (VISION)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200095-0022; 2015-005696-24 (EudraCT Number); 2024-512003-39-00 (EU CTIS Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-12 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced (Stage IIIB/IV) Non-small Cell Lung Cancer (NSCLC) With MET Exon 14 (METex14) Skipping Alterations or MET Amplification; Lung Adenocarcinoma Stage IIIB/IV
Keywords: lung; neoplasm; cancer; tumor; adenocarcinoma; MET exon 14; METex14; pulmonary; stage III; stage IV; c-Met; cMET; NSCLC; advanced non-small cell lung cancer; MET amplification; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Adenocarcinoma | interventions — tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1: Cohort A: METex14 Skipping Alterations (Other): Participants received 500 milligram (mg) of tepotinib once daily in cycles of 21-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Tepotinib
- Part 1: Cohort B: MET Amplification (Other): Participants received 500 milligram (mg) of tepotinib once daily in cycles of 21-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Tepotinib
- Part 2: Cohort C: Confirmatory Part for METex14 Skipping Alterations (Other): Participants received 500 milligram (mg) of tepotinib once daily in cycles of 21-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Subjects will receive 500 milligram (mg) of tepotinib once daily in cycles of 21-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.

SUMMARY:
This study looked at how effective the study drug (tepotinib) was at stopping the growth and spread of lung cancer. This study also measures a number of other things including safety of the study drug and the side effects, how body processes the study drug, or how the study drug affects your quality of life. The study also has an optional pharmacogenetic research part. Pharmacogenetic research is an important way to try to understand the role of genetics in human disease and how genes impact the effectiveness of drugs, because differences in genes can change the way a person responds to a particular drug.

DETAILED DESCRIPTION:
The study included 3 cohorts with one primary endpoint (Objective Response Rate). Enrollment number and completion data is changed by new cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent by participant or legal representative prior to any trial-specific screening procedure
* Male or female, greater than or equal to (>=) 18 years of age (or have reached the age of majority according to local laws and regulations)
* Measurable disease confirmed by an independent review committee (IRC) in accordance with RECIST version 1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* A female participant was eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential OR
* A woman of childbearing potential who agrees to use a highly effective contraception
* A male participant must agree to use and to have their female partners of childbearing potential to use a highly effective contraception
* Histologically or cytologically confirmed advanced (locally advanced or metastatic) NSCLC (all types including squamous and sarcomatoid)
* Treatment naïve participant in first-line or pretreated participant with no more than 2 lines of prior therapy
* Participants with MET alterations, namely METex14 skipping alterations in plasma and/or tissue as determined by the central laboratory or by an assay with appropriate regulatory status

Exclusion Criteria:

* Participants with characterized Epidermal Growth Factor Receptor (EGFR) activating mutations that predict sensitivity to anti-EGFR-therapy
* Participants with characterized Anaplastic Lymphoma Kinase (ALK) rearrangements that predict sensitivity to anti-ALK therapy
* Participants with symptomatic brain metastases who are neurologically unstable
* Any unresolved toxicity Grade 2 or more according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) from previous anticancer therapy
* Need for transfusion within 14 days prior to the first dose of trial treatment
* Prior chemotherapy, biological therapy, radiation therapy, hormonal therapy for anti-cancer purposes, targeted therapy, or other investigational anticancer therapy (not including palliative radiotherapy at focal sites) within 21 days prior to the first dose of trial treatment;
* Participants who have brain metastasis as the only measurable lesion
* Inadequate hematological, liver, renal, cardiac function
* Prior treatment with other agents targeting the Hepatocyte Growth Factor c(HGF/c) -Met pathway
* Hypertension uncontrolled by standard therapies (not stabilized to < 150/90 mmHg)
* Past or current history of neoplasm other than Non-small Cell Lung Cancer (NSCLC), except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer curatively treated and with no evidence of disease for at least 5 years
* Medical history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the test product
* Major surgery within 28 days prior to Day 1 of trial treatment
* Known infection with human immunodeficiency virus, or an active infection with hepatitis B or hepatitis C virus
* Substance abuse, active infection, or other acute or chronic medical or psychiatric condition or laboratory abnormalities that might increase the risk associated with trial participation at the discretion of Investigators
* Known hypersensitivity to any of the trial treatment ingredients
* Legal incapacity or limited legal capacity
* Any other reason that, in the opinion of the Principal Investigator, precludes the participant from participating in the trial
* Participation in another clinical trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc, a business of Merck KGaA, Darmstadt, Germany
Locations (167):
- United States (39):
  - City of Hope Cancer Center, Duarte, California
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - St. Joseph Hospital, Orange, California
  - Torrance Health Association, Redondo Beach, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Ingalls Hospital, Harvey, Illinois
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - For Recruiting Locations in the United States, please Contact U.S. Medical Information, Rockland, Massachusetts
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Summit Medical Group, P.A., Berkeley Heights, New Jersey
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Regional Cancer Care Associates East Brunswick, East Brunswick, New Jersey
  - Somerset Hematology Oncology Associates - Somerville Location, East Brunswick, New Jersey
  - Hackensack University Medical Center PARTNER, Hackensack, New Jersey
  - Prospect Medical Offices, LLC, Midland Park, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, West Harrison Regional Outpatient Pavilion, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - University of Cincinnati - PARENT, Cincinnati, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology, P.A. - Austin, Austin, Texas
  - Texas Oncology, PA, Beaumont, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Wenatchee Valley Hospital & Clinics - ATTN: Jay Johnson, Wenatchee, Washington
  - Wenatchee Valley Medical Center Oncology, Wenatchee, Washington
- LKH - Universitätsklinikum der PMU Salzburg - Innere Med III/Hämatologie und Onkologie, Salzburg, Austria
- Belgium (3):
  - UZ Antwerpen, Edegem
  - CHU Ambroise Paré, Mons
  - AZ Delta, Roeselare
- China (16):
  - Beijing Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital - Oncology, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Guangdong General Hospital, Guangzhou
  - Zhejiang Cancer Hospita, Hangzhou
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Cancer Hospital aka West Branch of Anhui Province Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Linyi Tumor Hospital, Linyi
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Cancer Hospital, Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The Affiliated Cancer Hospital of Xinjiang Medical university, Ürümqi
- France (22):
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac, Gironde
  - CHU de Toulouse - Hôpital Larrey, Toulouse, Haute Garonne
  - ICO - Site René Gauducheau, Saint-Herblain, Loire Atlantique
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire, Loire Atlantique
  - ICO - Site Paul Papin, Angers, Maine Et Loire
  - Centre Hospitalier de Cholet, Cholet, Maine Et Loire
  - Centre Hospitalier de Bretagne Sud, Lorient, Morbihan
  - Hopital Albert Calmette - CHU Lille, Lille, Nord
  - Centre Hospitalier de la côte Basque, Bayonne, Pyrenees Atlantiques
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon, Vendee
  - ICO - Site Paul Papin, Angers
  - Centre Hospitalier de la côte Basque, Bayonne
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Hopital Albert Calmette - CHU Lille, Lille
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Hôpital Saint-Louis, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac
  - ICO - Site René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (15):
  - POIS Leipzig GbR, Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Asklepios Fachkliniken Muenchen-Gauting, Gauting
  - SRH Wald-Klinikum Gera gGmbH, Gera
  - Universitaetsmedizin Goettingen, Göttingen
  - Evangelisches Krankenhaus Hamm GmbH, Hamm
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg / Saar
  - POIS Leipzig GbR, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Pius-Hospital Oldenburg, Oldenburg
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Ospedale Santa Maria di Cà Foncello, Padua
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Università Campus Bio-Medico di Roma, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (13):
  - NHO Kyushu Medical Center, Fukuoka
  - National Cancer Center Hospital East, Kashiwa-shi
  - Saitama Cancer Center, Kitaadachi-gun
  - Kurume University Hospital, Kurume-shi
  - NHO Shikoku Cancer Center, Matsuyama
  - Nagoya University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Sakaishi
  - Hokkaido University Hospital, Sapporo
  - NHO Yamaguchi - Ube Medical Center, Ube-shi
  - Kanagawa Cancer Center, Yokohama
  - Tottori University Hospital, Yonago-shi
- Netherlands (3):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG) - Parent, Groningen
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku - Dept of Pulmonology & Tuberculosis, Bialystok
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra
  - Dr n med. Slawomir Mandziuk Specjalistyczna Praktyka Lekarska, Lublin
  - NZOZ Olsztynski Osr. Onkologiczny "Kopernik" Sp.z o.o, Olsztyn
  - Przychodnia Med-Polonia Sp. z o.o., Poznan
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
- South Korea (12):
  - Dong-A University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (14):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona
  - Hospital General Universitario Santa Lucia, Cartagena
  - Hospital de Especialidades de Jerez de la Frontera - Servicio de Oncologia, Jerez de la Frontera
  - Hospital Universitario HM Madrid Sanchinarro, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern - Klinik und Poliklinik für Medizinische Onkologie, Bern
  - Universitaetsspital Zuerich - Klinik fuer Onkologie, Zurich
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Paik PK, Felip E, Veillon R, Sakai H, Cortot AB, Garassino MC, Mazieres J, Viteri S, Senellart H, Van Meerbeeck J, Raskin J, Reinmuth N, Conte P, Kowalski D, Cho BC, Patel JD, Horn L, Griesinger F, Han JY, Kim YC, Chang GC, Tsai CL, Yang JC, Chen YM, Smit EF, van der Wekken AJ, Kato T, Juraeva D, Stroh C, Bruns R, Straub J, Johne A, Scheele J, Heymach JV, Le X. Tepotinib in Non-Small-Cell Lung Cancer with MET Exon 14 Skipping Mutations. N Engl J Med. 2020 Sep 3;383(10):931-943. doi: 10.1056/NEJMoa2004407. Epub 2020 May 29. PMID 32469185
- [Derived] Kato T, Yang JC, Ahn MJ, Sakai H, Morise M, Chen YM, Han JY, Yang JJ, Zhao J, Hsia TC, Berghoff K, Bruns R, Vioix H, Lang S, Johne A, Le X, Paik PK. Efficacy and safety of tepotinib in Asian patients with advanced NSCLC with MET exon 14 skipping enrolled in VISION. Br J Cancer. 2024 Jun;130(10):1679-1686. doi: 10.1038/s41416-024-02615-9. Epub 2024 Apr 4. PMID 38575731
- [Derived] Le X, Paz-Ares LG, Van Meerbeeck J, Viteri S, Galvez CC, Smit EF, Garassino M, Veillon R, Baz DV, Pradera JF, Sereno M, Kozuki T, Kim YC, Yoo SS, Han JY, Kang JH, Son CH, Choi YJ, Stroh C, Juraeva D, Vioix H, Bruns R, Otto G, Johne A, Paik PK. Tepotinib in patients with non-small cell lung cancer with high-level MET amplification detected by liquid biopsy: VISION Cohort B. Cell Rep Med. 2023 Nov 21;4(11):101280. doi: 10.1016/j.xcrm.2023.101280. Epub 2023 Nov 8. PMID 37944528
- [Derived] Mazieres J, Paik PK, Garassino MC, Le X, Sakai H, Veillon R, Smit EF, Cortot AB, Raskin J, Viteri S, Wu YL, Yang JCH, Ahn MJ, Ma R, Zhao J, O'Brate A, Berghoff K, Bruns R, Otto G, Johne A, Felip E, Thomas M. Tepotinib Treatment in Patients With MET Exon 14-Skipping Non-Small Cell Lung Cancer: Long-term Follow-up of the VISION Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2023 Sep 1;9(9):1260-1266. doi: 10.1001/jamaoncol.2023.1962. PMID 37270698
- [Derived] Hallick J, Baird AM, Falchook G, Le X, Hong D, Viteri S, Raskin J, Reinmuth N, Vlassak S, Militaru M, Paik PK. Plain language summary of the development of tepotinib: a treatment for a subtype of non-small cell lung cancer called MET exon 14 skipping. Future Oncol. 2023 Mar;19(10):683-696. doi: 10.2217/fon-2022-1035. Epub 2023 Mar 31. PMID 36999526
- [Derived] Xiong W, Hietala SF, Nyberg J, Papasouliotis O, Johne A, Berghoff K, Goteti K, Dong J, Girard P, Venkatakrishnan K, Strotmann R. Exposure-response analyses for the MET inhibitor tepotinib including patients in the pivotal VISION trial: support for dosage recommendations. Cancer Chemother Pharmacol. 2022 Jul;90(1):53-69. doi: 10.1007/s00280-022-04441-3. Epub 2022 Jun 30. PMID 35771259
- [Derived] Xiong W, Papasouliotis O, Jonsson EN, Strotmann R, Girard P. Population pharmacokinetic analysis of tepotinib, an oral MET kinase inhibitor, including data from the VISION study. Cancer Chemother Pharmacol. 2022 May;89(5):655-669. doi: 10.1007/s00280-022-04423-5. Epub 2022 Apr 6. PMID 35385993
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095-0022
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Targeting MET Clinical Trial Program — https://www.clinicaltrials.targeting-met.com/en
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For Cohort A: A total of 168 participants were screened of which 152 participants were enrolled to receive the study drug. For Cohort B: A total of 32 participants were screened of which 24 participants were enrolled to receive the study drug. For Cohort C: A total of 175 participants were screened of which 161 participants were enrolled to receive the study drug.
Period: Overall Study
Arm/Group | Part 1: Cohort A: METex14 Skipping Alterations | Part 1: Cohort B: MET Amplification | Part 2: Cohort C: Confirmatory Part for METex14 Skipping Alterations
Started | 152 | 24 | 161
Completed | 137 | 23 | 128
Not Completed | 15 | 1 | 33
Not completed — still on treatment | 15 | 1 | 33

BASELINE CHARACTERISTICS:
Population: All participants in Cohort A, Cohort B and Cohort C who were administered at least 1 dose of tepotinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort A: METex14 Skipping Alterations | Part 1: Cohort B: MET Amplification | Part 2: Cohort C: Confirmatory Part for METex14 Skipping Alterations | Total
Number analyzed (Participants) | 152 | 24 | 161 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (8.97) | 62.3 (9.17) | 71.5 (9.24) | 71.5 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 3 | 86 | 162
  Male | 79 | 21 | 75 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 148 | 23 | 157 | 328
  Unknown or Not Reported | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 38 | 07 | 68 | 113
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 01 | 0 | 02 | 3
  White | 108 | 17 | 87 | 212
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 05 | 0 | 04 | 9

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Cohort A: Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Independent Review Committee (IRC)
Description: Objective response will be determined according to RECIST 1.1 and as per IRC. Objective response was defined as number of participants with either a confirmed complete response (CR) or partial response (PR) from first administration of study treatment to first observation of progressive disease (PD) .CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first treatment up to data cutoff (approximately Month 66)
Population: Safty Analysis Set included all participants in Cohort A who were administered at least 1 dose of tepotinib, including participants with METex14 skipping alterations not confirmed by a validated central laboratory assay.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A: METex14 Skipping Alterations
Number analyzed (Participants) | 152
percentage of participants | 46.7 [38.6 to 55.0]

2. Primary Outcome: Part 1: Cohort B: Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 as Assessed by Independent Review Committee (IRC)
Description: as for outcome 1
Time Frame: Time from first treatment up to data cutoff (approximately Month 66)
Population: Safety Analysis Set included all participants in Cohort B who were administered at least 1 dose of tepotinib, including participants with a MET Amplification.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort B: MET Amplification
Number analyzed (Participants) | 24
percentage of participants | 41.7 [22.1 to 63.4]

3. Primary Outcome: Part 2: Cohort C: Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 as Assessed by Independent Review Committee (IRC)
Description: as for outcome 1
Time Frame: Time from first treatment up to data cutoff (approximately Month 66)
Population: Safety analysis set included all participants in Cohort C who were administered at least 1 dose of tepotinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Cohort C: Confirmatory Part for METex14 Skipping Alterations
Number analyzed (Participants) | 161
percentage of participants | 54.7 [46.6 to 62.5]

4. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Duration of Response (DOR) Assessed by Investigator
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

6. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Duration of Response (DOR) Assessed by Investigator
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

7. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Objective Disease Control Rate Assessed by IRC
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

8. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Objective Disease Control Rate Assessed by Investigator
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

9. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Progression-free Survival by IRC Assessment
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

10. Secondary Outcome: Part 1 & 2: Cohort A + B +C: Progression-free Survival by Investigator Assessment
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

11. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Overall Survival (OS)
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

12. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

13. Secondary Outcome: Part 1 & 2: Cohort A + B +C: Number of Participants With Markedly Abnormal Clinical Laboratory Tests
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

14. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Number of Participants With Markedly Abnormal Vital Signs and Physical Examination
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

15. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Number of Participants With Clinically Significant Change From Baseline in 12-Lead Electrocardiogram (ECG)
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

16. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Change From Baseline in Euro Quality of Life Questionnaire With 5 Questions Alternatives (EQ5D-5L) Summary Score
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

17. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

18. Secondary Outcome: Part 1 & 2: Cohort A + B + C: Quality of Life (QoL) Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Time Frame: Time from first treatment up to end of study (approximately Month 101)
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Time from first treatment up to data cutoff (approximately Month 74)
Groups:
- Part 1 & 2: Cohort A + B + C: Participants received 500 milligram (mg) of tepotinib once daily in cycles of 21-day duration until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
Arm/Group | Part 1 & 2: Cohort A + B + C
All-Cause Mortality (participants affected / at risk) | 200/337
Serious Adverse Events (participants affected / at risk) | 169/337
Other Adverse Events (participants affected / at risk) | 331/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 & 2: Cohort A + B + C (N=337)
Anaemia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myopericarditis (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chest pain (General disorders) | 1
Death (General disorders) | 2
Disease progression (General disorders) | 16
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 12
Generalised oedema (General disorders) | 8
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 11
Pyrexia (General disorders) | 3
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Bacterial infection (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Pleural infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 18
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic embolus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Urinary tract infection bacterial (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Troponin increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aphasia (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 3
Vocal cord paresis (Nervous system disorders) | 1
Stent malfunction (Product Issues) | 1
Assisted suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Delusion (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 & 2: Cohort A + B + C (N=337)
Anaemia (Blood and lymphatic system disorders) | 50
Lacrimation increased (Eye disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 29
Abdominal pain upper (Gastrointestinal disorders) | 29
Constipation (Gastrointestinal disorders) | 69
Diarrhoea (Gastrointestinal disorders) | 95
Nausea (Gastrointestinal disorders) | 97
Vomiting (Gastrointestinal disorders) | 46
Asthenia (General disorders) | 46
Fatigue (General disorders) | 51
Generalised oedema (General disorders) | 22
Oedema (General disorders) | 31
Oedema peripheral (General disorders) | 237
Pyrexia (General disorders) | 33
Pneumonia (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 23
Fall (Injury, poisoning and procedural complications) | 18
Alanine aminotransferase increased (Investigations) | 56
Amylase increased (Investigations) | 34
Aspartate aminotransferase increased (Investigations) | 40
Blood alkaline phosphatase increased (Investigations) | 35
Blood creatinine increased (Investigations) | 96
Gamma-glutamyltransferase increased (Investigations) | 28
Lipase increased (Investigations) | 28
Weight decreased (Investigations) | 22
Decreased appetite (Metabolism and nutrition disorders) | 65
Hypoalbuminaemia (Metabolism and nutrition disorders) | 108
Hypocalcaemia (Metabolism and nutrition disorders) | 33
Hypokalaemia (Metabolism and nutrition disorders) | 25
Hyponatraemia (Metabolism and nutrition disorders) | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 69
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 37
Alopecia (Skin and subcutaneous tissue disorders) | 36
Dry skin (Skin and subcutaneous tissue disorders) | 30
Pruritus (Skin and subcutaneous tissue disorders) | 26
Rash (Skin and subcutaneous tissue disorders) | 30
Hypotension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02864992/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02864992/SAP_001.pdf